CLINICAL TRIAL: NCT01458093
Title: Large Overuse of Post-polypectomy Surveillance Colonoscopy: a Prospective Nation-wide Study
Brief Title: Large Overuse of Post-polypectomy Surveillance Colonoscopy
Status: Completed | Type: Observational
Sponsor: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Franco Radaelli, Principal Investigator, Valduce Hospital
Other Study IDs: SURV_2011
Record Dates: First submitted 2011-10-18; First posted 2011-10-24 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Colonic Polyps; Surveillance; Colonoscopy
MeSH Terms: conditions — Colonic Polyps | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Colonoscopy patients: Consecutive colonoscopy outpatients referred to one of 29 endoscopy units in Italy
  Interventions: Other: colonoscopy

INTERVENTIONS:
Other: colonoscopy — evaluation of surveillance timing adequacy as compared to the guidelines

SUMMARY:
In colorectal cancer screening era a huge burden of medical resources has been applied to surveillance. Although the adherence to post-polipectomy recommendations is a advocated as a mainstay for quality assurance colonoscopy programs, prospective data on appropriateness of surveillance are lacking.

The aim of present study was to evaluate the percentage of subjects in which timing of surveillance colonoscopy in practice agrees with that recommended by guidelines and to identify factors associated to the appropriateness of surveillance.

ELIGIBILITY:
Inclusion Criteria:

* consecutive colonoscopy outpatients
* adults (18-80 yrs)

Exclusion Criteria:

* Subjects with missing data on polyp findings at previous colonoscopy (number, endoscopic or histological features)
* Subjects with unsatisfactory quality standards of previous examination (no cecal intubation, inadequate bowel preparation, incomplete polyp resection)
* patients with a medical history of inflammatory bowel disease, inherited or other polyposis syndrome and colorectal cancer.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred to one out of 29 endoscopy units in Italy to undergo colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 7081 (Actual)
Dates: Start 2010-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Adherence to post-polypectomy surveillance guidelines | up to one year
  Time interval between index and surveillance colonoscopies for patients undergoing post-polypectomy surveillance was calculated and compared to that suggested by the guidelines according to endoscopic findings at previous examination. For each patiens, surveillance time interval was regarded as correct if coherent with the recommended interval +/- 6 months, thus allowing to calculate the proportion of correct prescriptions

SECONDARY OUTCOMES:
Factors associated to surveillance appropriateness | up to one year
  The presence of factors associated to appropriate surveillance prescriptions was investigated by multivariate analysis (odds ratio and 95% confidence interval for each factor)

CONTACTS AND LOCATIONS:
Locations (1):
- Valduce Hospital, Como, Italy

REFERENCES:
- [Derived] Radaelli F, Paggi S, Bortoli A, De Pretis G; Italian Association of Hospital Gastroenterologists (AIGO). Overutilization of post-polypectomy surveillance colonoscopy in clinical practice: a prospective, multicentre study. Dig Liver Dis. 2012 Sep;44(9):748-53. doi: 10.1016/j.dld.2012.04.015. Epub 2012 May 22. PMID 22627070